CLINICAL TRIAL: NCT01283711
Title: Evaluation of Safety and Efficacy of the Apollo™ System for Treatment of Wrinkles and Rhytides
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pollogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC210114_A
Record Dates: First submitted 2011-01-25; First posted 2011-01-26 (Estimated); Last update posted 2013-05-17 (Estimated); Status verified 2011-11

CONDITIONS: Facelift
Keywords: wrinkles reduction; rhytides reduction; RF treatment

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- apollo (Experimental)
  Interventions: Device: apollo device

INTERVENTIONS:
Device: apollo device — RF treatments for wrinkles and rhytides reduction

SUMMARY:
Non-invasive, energy-based, aesthetic treatments are becoming increasingly popular among female and male patients of all ages. Different technologies are presently available to rejuvenate skin, including therapeutic ultrasound, lasers and intense pulsed light (IPL), however radiofrequency has emerged as the most effective and versatile modality for the broadest range of body and facial treatments, including non-invasive wrinkle treatment.

The apollo™ system is an RF system, based on the TriPollar™ technology. The technology is based on three or more electrodes designed to deliver RF current focused into the skin, thus generating heat in the dermal layer. Selective and focused electro-heating of the skin is intended to stimulate collagen remodeling in the dermal layer resulting in non invasive wrinkle treatment.

The apollo™ system is intended for use in dermatologic and general surgical procedures for non invasive treatment of facial wrinkles and rhytides. This study was designed in order to evaluate the safety and efficacy of the Apollo™ System for facial wrinkles and rhytides treatments.

ELIGIBILITY:
Inclusion Criteria:

* Subject read, understood and signed the Consent Form
* Healthy female/male aged 35 65 years,
* Fitzpatrick wrinkle classification score 4 and above
* Subject is capable of reading, understanding and following instructions of the procedure to be applied.
* Subject is able and willing to comply with the treatment and follow-up schedule.

Exclusion Criteria:

* Subject has a pacemaker or internal defibrillator, implanted neurostimulators or any other internal electric device or patient who had an implant in the past.
* Subject has metal or other implants in the treatment area (Not including dental fillings, implants and crowns).
* Subject has current or history of cancer, especially skin cancer or premalignant moles or is undergoing any form of treatment for active cancer.
* Subject has severe concurrent conditions such as epilepsy, lupus or cardiac disorders.
* Subject has poorly controlled endocrine disorders such as diabetes.
* Subject is female who is pregnant, lactating, or plans to become pregnant during the study period or had given birth less than 6 months ago.
* Subject has an impaired immune system due to immunosuppressive diseases such as HIV or AIDS, or use of immunosuppressive medications.
* Subject has a condition that could be negatively affected by heat, including any history of diseases stimulated by heat, such as recurrent Herpes Simplex (in the treatment area).
* Subject has diminished or exaggerated perception of temperature changes.
* Subject has significant concurrent skin conditions affecting areas to be treated such as sores, hemorrhages or risk of hemorrhages, septic conditions, psoriasis, eczema and rash as well as very dry and fragile skin.
* Subject has history of collagen disorders, keloid formation and abnormal wound healing.
* Subject has had previous invasive/ablative procedures in the areas to be treated within 3 months prior to initial treatment or plans on such treatment during the course of the study, or before complete healing has occurred.
* Subject has had Botox injections in the treatment area within 6 months prior to initial treatment
* Subject has had natural fillers within 9 months prior to initial treatment
* Subject has synthetic fillers or gold/plastic threads in the treatment area.
* Subject takes or has taken medications, herbal preparations, food supplements or vitamins that might cause fragile skin or impaired skin healing such as prolonged steroid regime, tetracyclines, or St. John's Wort for the last 3 months.
* Subject has used oral isotretinoin (Accutane or Roaccutan) within 6 months prior to study enrollment or plans use during the course of the study.
* Subject has history of bleeding coagulopathies or use of anticoagulants.
* Subject has burned, blistered, irritated, or sensitive skin due to excessive fresh tanning in areas to be treated or is unlikely to refrain from excessive tanning during the study.
* Concurrent participation in any other study.
* Subject has mental disorders.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2011-03; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety of the apollo™ system for wrinkles and rhytides treatment. | 5 months
  The safety of using the apollo™ system for wrinkles and rhytides treatment will be established by physician's assessment/observation of adverse events.

SECONDARY OUTCOMES:
• To evaluate the efficacy of the apollo™ system for wrinkles and rhytides treatment. | 5 months
  Efficacy of using the apollo™ system for wrinkles and rhytides treatment will be established by level of wrinkle reduction.

CONTACTS AND LOCATIONS:
Overall Officials: Mira Barki, Dr., Study Director — Pollogen
Locations (2):
- Steven D. Shapiro MD, Palm Beach Gardens, Florida, United States
- Kaplan Medical center, Rehovot, Israel